CLINICAL TRIAL: NCT05357599
Title: The Use of Endoscopic Ultrasound-Guided Portal Pressure Measurements to Guide Beta-Blocker Therapy in Patients With Compensated Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, James Buxbaum, Chief of Gastroenterology Los Angeles County + University of Southern California, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APP-22-01828
Record Dates: First submitted 2022-04-17; First posted 2022-05-03 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Cirrhosis; Compensated Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Fibrosis; Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Beta Blocker at EUS (Experimental)
  Interventions: Diagnostic Test: EUS

INTERVENTIONS:
Diagnostic Test: EUS — The decision to start a beta-blocker will be made at the conclusion of the EGD based on the endoscopic findings (presence of esophageal varices)

SUMMARY:
This pilot study to determine the feasibility of EUS-Portal Pressure Measurements to guide Beta-Blocker Therapy in patients with compensated cirrhosis .The study will be a prospective tandem controlled trial consisting of 30 patients who are already undergoing routine endoscopy screening for portal hypertension as part of their routine clinical care . The decision to start a beta-blocker will be made at the conclusion of the EGD based on the endoscopic findings (presence of esophageal varices). EUS-PPG will then be performed and measurements will be collected. The primary outcome is the feasibility of guiding B blocker therapy by EGD+EUS-PPG at the time of EGD for variceal screening. The secondary outcome will be the proportion of patients initiated on beta-blocker therapy based on EGD alone versus EGD+EUS-PPG

DETAILED DESCRIPTION:
The study will be a prospective tandem controlled trial consisting of 30 patients who are undergoing EGD followed by EUS-PPG at Los Angeles County + University of Southern California Medical Center (LAC+USC).

Only patients undergoing endoscopic screening for portal hypertension as part of routine clinical care will be considered for the study.

All procedures will be performed with the patient under moderate sedation or monitored anesthesia care as is standard in our endoscopy unit. EGD with a forward-viewing scope will be performed initially in all patients to evaluate and document the presence of esophageal varices. Any other endoscopic evidence of portal hypertension, such as portal hypertensive gastropathy or gastric varices, will also be documented.

The decision to start a beta-blocker will be made at the conclusion of the EGD based on the endoscopic findings (presence of any esophageal varices).

EUS-PPG will then be performed. Using the dedicated 25-gauge portal systemic pressure measurement needle, the hepatic venous system and portal venous system will be directly accessed to allow measurements. The mean portal pressure gradient will be recorded. We will then record whether beta-blockers would be initiated based on portal pressure measurements ≥10mmHg.

The peri-procedure management will be performed according to standard of care within our endoscopy unit. As is our standard clinical care for patients with portal hypertension, for patients found to have evidence of portal hypertension we will start the beta-blocker carvedilol 6.25mg twice a day will be started on the day following the procedure. If tolerated, the dose will be increased to 12.5mg twice a day after one month.

The patients will be blinded to whether or not the decision to start beta-blockers was based on EGD, EUS-PPG or both findings. The patient will be followed clinically by the principal investigator assisted by a full time study coordinator and team with extensive prospective clinical trials experience

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age.
2. diagnosis of Child-Pugh class A cirrhosis who present to LAC+USC for variceal screening.

A diagnosis of cirrhosis will be determined histologically based on biopsy alone or clinically by reviewing notes from a gastroenterology or hepatology provider with imaging and clinical history consistent with cirrhosis.

Exclusion Criteria:

1. Prior decompensation, which includes a history of variceal hemorrhage, ascites, and/or hepatic encephalopathy;
2. other complications of cirrhosis that can affect portal pressures, such as splenic or portal vein thrombosis and/or hepatocellular carcinoma,
3. use of any medications (i.e. current beta-blocker use) or prior procedure that affects splanchnic hemodynamics or portal pressure;
4. contraindications to beta-blockers, including resting heart rate <60, systolic blood pressure <90, history of bronchospasm;
5. current incarceration;
6. pregnancy; and
7. inability to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of guiding B blocker therapy for variceal screening | Procedure through study completion, an average of 7 days
  Feasibility will be measured by procedure success, Intra-procedure times, and adverse events.

SECONDARY OUTCOMES:
Initiation on beta-blocker therapy based EGD alone versus EGD+EUS-PPG. | Baseline
  The secondary outcome will be the proportion of patients initiated on beta-blocker therapy based on EGD alone versus EGD+EUS-PPG.

CONTACTS AND LOCATIONS:
Overall Officials: James Buxbaum, MD, Principal Investigator — LAC+USC Medical Center

IPD SHARING:
Plan to Share IPD: Undecided